CLINICAL TRIAL: NCT03727165
Title: Cyclic Enteral Nutrition Versus Continuous Infusion of Enteral Nutrition in Achieving Caloric Goals: Randomized Clinical Trial
Brief Title: Nocturnal Cyclic Enteral Nutrition Infusion Versus Continuous Infusion of Enteral Nutrition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid pandemia.suspended study
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/121
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Critical Illness; Enteral Feeding Intolerance; Nutrition Support
Keywords: enteral nutrition; critically ill; continous infusion; cyclic infusion
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be in the intensive care unit under sedative treatment and will not know about randomization Nurses in the intensive care unit (care providers of enteral nutrition infusion) will not know about the study Outcomes evaluation will be made by one independent clinical epidemiologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous infusion (Active Comparator): Patients with continuous infusion enteral nutrition in the intensive care unit at San Ignacio University Hospital
  Interventions: Other: Continuous enteral nutrition infusion
- Cyclic infusion (Experimental): Patients formulated with cyclic enteral nutrition infusion, administrated at night hours, from 4pm until 7am.
  Interventions: Other: Cyclic enteral nutrition infusion

INTERVENTIONS:
Other: Continuous enteral nutrition infusion — Enteral nutrition administration in continuous infusion during 24 hours per day
  Arms: Continuous infusion
Other: Cyclic enteral nutrition infusion — Enteral nutrition administration in continuous infusion during 16 hours per day
  Arms: Cyclic infusion

SUMMARY:
Enteral nutrition is considered the best way to feed those who can´t be fed orally. the standard protocol of administration includes continuous infusion for 24 hours; nonetheless this support is constantly suspended which causes a decrease in the nutrition administered vs the one formulated.

Therefore this randomized clinical trial attempts to compare de standard administration vs. cyclic infusion during night hours measuring the formulated vs the administered volume of enteral nutrition given to the patient.

The control group will be assigned standard 24 hour infusion of enteral nutrition while the experimental group will be assigned cyclic infusion during night hours. The variables include volume formulated, volume given in 24 hours, hours and reasons why the enteral nutrition was suspended, and related complications (abdominal distension, vomiting, and diarrhea).

DETAILED DESCRIPTION:
The trial will be carried at San Ignacio University Hospital intensive care unit. Patients included will be over 18 years old who require enteral nutrition according to their attending or to the nutritional and metabolic support team.

260 envelopes with the specific intervention were created. 130 of them are identified with number 0 which corresponds to no intervention, meaning continuous enteral nutrition infusion during 24 hours. The other 130 are assigned with the number 1 which corresponds to intervention, meaning nocturnal cyclic nocturnal enteral nutrition infusion.

Envelopes will be randomly assigned sequentially from number 1 to 260, in which envelope number 1 will be assigned for the first patient. Each patient´s envelope will be labeled with its name and identification number. According to the information contained in the envelope the specific scheme assigned will be formulated.

Envelopes will be kept at the Nutritional and metabolic support´s office; only research assistant will have access to this information.

After 50% of the sample be achieved, there will be a data analysis to review the rate of intolerance to enteral nutrition in both groups.

Principal investigators will review the entire data after completion of the clinical trial, measuring percentage of enteral nutrition delivered and intolerance to enteral nutrition feeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, hospitalized in San Ignacio University Hospital intensive care unit.
* Patients with indication on enteral nutrition defined by its attending or by the Nutritional and Metabolic support team.

Exclusion Criteria:

-If patient or legal advocate denies to sign consent to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Enteral nutrition delivered/Enteral nutrition prescribed x 100 | 24 hours
  Enteral nutrition delivered/Enteral nutrition prescribed x 100

SECONDARY OUTCOMES:
Enteral nutrition intolerance | 24 hours
  number of patients with intolerance/total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Saul J Rugeles, MD, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Bogota DC, Colombia

IPD SHARING:
Plan to Share IPD: No